CLINICAL TRIAL: NCT06589648
Title: The Effect of Mandala Coloring on Anxiety and Mental Fatigue Levels in Pregnant Women Diagnosed With Threatened Preterm Labor: A Randomized Controlled Trial
Brief Title: The Effect of Mandala Coloring on Anxiety and Mental Fatigue in Pregnant Women Diagnosed With Threatened Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Cennet Nur Bircan, Chief Researcher, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KTO- Midwifery- C.N.Bircan-001
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Anxiety During Pregnancy; Mental Fatigue; Mandala
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Intervention Model Description: mandala coloring
Who Masked: Participant, Outcomes Assessor
Masking Description: The research statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in the intervention group will be given a set of colored markers and a mandala coloring page and will be asked to color them any time of the day and in any way they want during their hospital stay. Participants will be asked to take a picture of the mandala they colored and send it to the researcher after they are finished. Participants will be reminded daily so that they do not forget to do the activity.
  Interventions: Other: mandala painting
- control group (No Intervention): No intervention other than routine care will be made to the control group of the study, and research data will be collected at simultaneous intervals with the experimental group.

INTERVENTIONS:
Other: mandala painting — Mandala coloring creates a relaxing effect on individuals because it starts with a pattern that develops like a flower around a point; it allows the individual to stay in the moment, to get away from stress, anxiety and worries, and it relaxes the mind.
  Arms: intervention group

SUMMARY:
The research will be conducted in a pre-test-post-test control group randomized control design. The aim is to examine the effect of mandala work on anxiety and mental fatigue in pregnant women diagnosed with threatened preterm labor. Hypotheses

1. Mandala coloring work reduces the level of anxiety related to pregnancy in pregnant women diagnosed with threatened preterm labor.
2. Mandala coloring work reduces the level of anxiety in pregnant women diagnosed with threatened preterm labor.
3. Mandala coloring work reduces the level of mental fatigue in pregnant women diagnosed with threatened preterm labor.

Pregnant women who meet the inclusion criteria will be given general information about the research before randomization, their consent will be obtained and pre-test data will be collected. Pregnant women whose pre-test data are collected will be assigned to the intervention and control groups using the simple randomization method.

Intervention group: Participants in the intervention group will be given a set of colored markers and a mandala coloring page and will be asked to color them at any time of the day and in any way they want during their hospitalization. Participants will be asked to take a picture of the mandala they colored and send it to the researcher after they are finished. Participants will be reminded daily so that they do not forget to do the activity. Research data will be collected a total of four times before randomization, on the 1st day, 2nd day and 3rd day after the mandala application was started.

Control Group: No intervention other than routine care will be made to the control group of the study, and research data will be collected at simultaneous time intervals with the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who can read and write Turkish,
* Diagnosed with threatened preterm labor,
* Are between 32-36 weeks of gestation,
* Primiparous,
* Hospitalized,
* Open to communication (able to understand and answer questions) will be included in the sample.

Exclusion Criteria:

* Pregnant women with a history of miscarriage or stillbirth,
* Those who voluntarily withdrew from the study,
* Those with a history of psychiatric illness (self-report),
* Those who do not have a physical disability that would prevent them from coloring mandalas will be excluded from the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Pregnancy-Related Anxiety Scale | 0-3 day
  It was developed by Brunton et al. (2019), which can be applied to primiparous and multiparous pregnant women, and adapted into Turkish by Şolt and Kanza Gül (2020). The scale is a 4-point Likert-type scale with 9 sub-dimensions: "Birth-Related Anxiety" (items 1, 2, 3, 4, 5, and 6), "Body Image Anxiety" (items 7, 8, 9, 10, and 11), "Attitudes Towards Birth" (items 12, 13, 14), "Concerns About Motherhood" (items 15, 16, 17), "Acceptance of Pregnancy" (items 18, 19, 20), "Anxiety Indicators" (items 21, 22, 23, and 24), "Attitudes Towards Healthcare Personnel" (items 25, 26, and 27), "Avoidance" (items 28, 29, and 30) and "Attitudes Towards the Baby" (items 29, 30, and 40). It consists of a total of 33 items, including "Anxiety" (items 31, 32 and 33). The lowest score is 33 and the highest is 132, and there is no cut-off point. As the scores obtained from the scale increase, anxiety related to pregnancy increases. The Cronbach Alpha coefficient of the scale was stated as 0.82 for multipa

SECONDARY OUTCOMES:
State Anxiety Inventory | 0-3 day
  It is a scale consisting of 20 questions developed by Speilberger et al. (1983) (Öner, 1997; Öner & Le Compte, 1985). It was adapted to Turkish by Öner and Le Compte (1974-1977) (Öner, 1997; Öner & Le Compte, 1985). The emotions or behaviors expressed in the items of the scale consist of the following options according to the severity of the experience: 1) Not at all, 2) A little, 3) A lot, and 4) Completely. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 of the scale are reverse-coded. The total score obtained from the scale varies between 20 and 80 (Öner, 1997; Öner & Le Compte, 1985). A high score indicates a high level of anxiety, a low score indicates a low level of anxiety.

OTHER OUTCOMES:
Mental Fatigue Scale | 0-3 day
  It is a multidimensional questionnaire consisting of 15 questions designed by Johansson et al. (2010). The scale covers sleep, sensory, emotional and cognitive areas, mental recovery and 24-hour changes. The cut-off score of the original scale was determined as 10.5. A score above this score indicates a problem, although not always serious (Johansson et al., 2010). The Turkish validity and reliability study of the scale with nurses was conducted by Güven et al. (2023) and mental fatigue states were assessed with 12 items. The questions include general fatigue, lack of initiative, mental fatigue, mental recovery, concentration difficulties, memory problems, slowness in thinking, sensitivity to stress, increased tendency to become emotional, irritability, sensitivity to light and noise, decreased or increased sleep, and 24-hour changes in symptoms. Each question has 4 descriptive rating options (0-3).

CONTACTS AND LOCATIONS:
Overall Officials: Karakoç, Study Director — KTO Karatay Univeristy
Locations (1):
- Necmettin Erbakan University Medical Faculty Hospital, Konya, Konya/ Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol